CLINICAL TRIAL: NCT01997242
Title: A Multicenter Registry of Consecutive Patients Undergoing Cardiac and Noncardiac Surgery or Operative Endoscopic/Endovascular Procedures After Implantation of a Coronary Stent
Brief Title: The Surgery After Stenting (SAS) Registry
Acronym: SAS registry
Status: Completed | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Collaborators: Italian Society of Invasive Cardiology (Other); Associazione Nazionale Medici Cardiologi Ospedalieri (Other)
Responsible Party: Sponsor
Other Study IDs: ASMN-18/2013
Record Dates: First submitted 2013-09-14; First posted 2013-11-28 (Estimated); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: PERCUTANEOUS CORONARY INTERVENTION; STENTS; SURGERY
Keywords: CORONARY STENT; CARDIAC SURGERY; NON CARDIAC SURGEY

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- stenting undergoing surgery: Patients with prior coronary stenting undergoing urgent or elective surgical/endoscopic procedures

SUMMARY:
The SAS registry will include any patient with previous coronary stenting undergoing any type of surgery or operative endoscopic/endovascular procedure at the participating Centers. The relevant clinical, procedural and outcome data (within index surgical admission and at 30 days) will be entered in a specifically designed electronic case record form (eCRF).

ELIGIBILITY:
Inclusion Criteria:

* Eligible will be male and female patients > 18 years of age.
* Eligible will be patients with previous coronary stenting undergoing any kind of surgical or operative endoscopic procedure at the participating Centers, irrespective of the distance in time between stenting and surgery.
* Both candidates to elective/urgent operations and those undergoing emergency operations will be included in the SAS registry, and will be considered as two separate cohorts.

Exclusion Criteria:

- Unwillingess/inability to sign the Informed Consent Form (ICF). There are no other selection criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with prior coronary stenting undergoing urgent or elective surgical/endoscopic procedures
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-06-10 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
The composite of death, myocardial infarction, probable/definite stent thrombosis according the Academic Research Consortium definition and bleeding events of Bleeding Academic Research Consortium (BARC)grade >3 during index surgical admission. | within the first 30 days after surgery

SECONDARY OUTCOMES:
The incidence of bleeding events of Bleeding Academic Research Consortium (BARC) grade >3 within 30 days of index admission/procedure | within the first 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Savonitto, MD, Study Chair — Division of Cardiology, Manzoni Hospital, Lecco; Roberta Rossini, MD, Study Chair — Cardiovascular Dpt, Ospedali Riuniti di Bergamo; Giovanni Tortorella, MD, Study Chair — Arcispedale Santa Maria Nuova - IRCCS, Reggio Emilia; Marco Ferri, MD, Principal Investigator — Arcispedale Santa Maria Nuova - IRCCS, Reggio Emilia
Locations (1):
- Arcispedale Santa Maria Nuova- IRCCS, Reggio Emilia, Italy, Italy